CLINICAL TRIAL: NCT00758849
Title: A Phase II, Randomised, Placebo-Controlled, Double-Blind, Replicated Crossover, Pilot Study on the Effect of Fipamezole on Neurogenic Orthostatic Hypotension in Patients With Multiple System Atrophy or Parkinson's Disease
Brief Title: Fipamezole in Neurogenic Orthostatic Hypotension
Acronym: Foehn
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Juvantia Pharma Ltd (Industry)
Collaborators: Santhera Pharmaceuticals (Industry)
Responsible Party: Juha M. Savola, Director Clinical Development, Santhera Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-II-005
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension (NOH); Parkinson's Disease; Multiple System Atrophy
Keywords: NOH; Orthostatic hypotension; PAF; MSA; Shy-Drager syndrome; Olivopontocerebellar atrophy; Striatonigral degeneration; Autonomic Failure; Parkinson; Fipamezole; JP-1730
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Hypotension, Orthostatic; Shy-Drager Syndrome; Olivopontocerebellar Atrophies; Striatonigral Degeneration; Pure Autonomic Failure | interventions — fipamezole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Fipamezole

INTERVENTIONS:
Drug: Placebo — One placebo tablet administered tid for 12 days in each of the three crossover treatment blocks, each block separated by 2-days placebo washout
  Arms: 1
Drug: Fipamezole — One 30-mg tablet of Fipamezole tid from day 1 to 3; one 60-mg tablet of Fipamezole tid from Day 4 to 6; and one 90-mg tablet of Fipamezole tid from Day 7 to 12 in each of the three crossover treatment blocks, each block separated by 2-days placebo washout
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Fipamezole is effective in the treatment of orthostatic hypotension and related symptoms in multiple system atrophy and Parkinson's disease.

DETAILED DESCRIPTION:
This study will be an exploratory, proof of concept, randomised, placebo-controlled, double-blind, multiple crossover study, with an open-label active run-in phase, in patients with multiple system atrophy (MSA) or Parkinson's disease (PD) who can concomitantly be treated with fludrocortisone and antiparkinsonian medication. Three sites in France and one site in Portugal will participate in this study.

During the open-label active run-in phase, a tolerated dose-escalation regimen (either escalating from 30 to 90 or 60 mg tid, or no escalation but fixed dose of 30 mg tid) will be established for each patient. Once the tolerated treatment regimen has been established, patients will then be randomised to the double-blind crossover treatment. Fipamezole and matched placebo tablets are compared in 3 crossover blocks, each block consisting of a total of 28 days: 12 days fipamezole and 12 days placebo in random order, separated by two days of washout. The patients will be randomly assigned to one of the two possible treatment sequences (fipamezole first followed by placebo or placebo first followed by fipamezole).

For efficacy assessments, the patient blood pressure and heart rate is assessed repeatedly when laying still or standing. Impact of orthostatic hypotension on clinical symptoms is assessed with a subjective scale and questionnaire. To explore potential positive or negative impact of fipamezole on disease characteristics, the MSA and PD patients are assessed with UMSARS and UPDRS scales, respectively. Finally, the study includes investigator and patients assessments of CGI-I and PGI-I scales for clinical condition in general.

Fipamezole

Fipamezole is a new antagonist of the pre-synaptic adrenergic alpha-2 receptors and is being investigated for potential use as an adjunctive therapy for PD. Adrenergic alpha-2 receptors inhibit noradrenaline and some other neurotransmitter release from nerve terminals in a tonic manner, and therefore antagonism of this receptor leads in enhanced neurotransmitter release. Alpha-2 receptors are located widely in the body, both in the central nervous system (CNS) and periphery. Pharmacological studies have suggested that either central or peripheral autonomic nervous system is involved in autonomic failure and orthostatic hypotension in MSA and in PD. Neurogenic orthostatic hypotension in these diseases results from decreased delivery of the sympathetic neurotransmitter noradrenaline (or hormonal adrenaline) to vascular adrenergic receptors, either because of blunted CNS control or impaired function of postganglionic sympathetic neurons. Fipamezole is expected to increase noradrenergic (or adrenergic) turnover in specific areas of the brain or in the periphery in MSA and PD and alleviate symptoms related to fall in BP during orthostatism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 30 and < 80 years of age with an intact oral mucosa at screening
* Diagnosis of MSA or diagnosis of idiopathic PD
* Hoehn and Yahr stages 1 to 4 during 'Off' period
* NOH: reproducible fall in SBP ≥20 mmHg and/or a fall in DBP ≥10 mmHg between 15 min of supine rest and 3 min of standing (or until symptomatic from hypotension after <3 min of standing)
* For patient taking antiparkinsonian medication: stable daily dosing for at least 1 month
* For patient taking fludrocortisone: stable dose for at least 2 months
* Demonstrated ability to comprehend, give informed consent and comply with study procedures (BP self-monitoring, completion of patient diary and self-assessment rating scales)

Exclusion Criteria:

* Other clinically significant conditions apart from those typically associated with MSA or PD
* SBP ≥200 mmHg or DBP ≥120 mmHg after 15 min supine rest in quiet environment
* Clinically significant abnormalities of ECG
* Mini-Mental State Examination (MMSE) score < 24
* Intake of prohibited concomitant medication such as midodrine, intake of medication associated with vasodilatation or induction of liver enzymes; neuroleptics; certain drugs known to be substantially metabolized through the following cytochrome P450 isoenzymes: 1A2, 2B6, 2C19, 2C9, 2D6 and 2E1; or any other drug for the treatment of orthostatic hypotension (including off-label use), such as non-steroidal anti-inflammatory drugs, beta blockers, somatostatin
* Use of St. John's Wort or Ginkgo Biloba within 48 h prior to inclusion and during the course of the study
* Intake of an investigational drug within 30 days prior to screening

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of fipamezole with that of placebo on orthostatic hypotension as assessed by blood pressure response to orthostatism. | 28 days

SECONDARY OUTCOMES:
To compare the efficacy of fipamezole with that of placebo on heart rate (HR) response to orthostatism. | 28 days
To compare the efficacy of fipamezole with that of placebo on clinical symptoms. | 28 days
To explore the relationship between plasma levels of fipamezole and measures of efficacy and safety (pharmacokinetics). | 28 days
To assess safety and tolerability of fipamezole. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rascol, MD, Principal Investigator — Hôpital Purpan CIC du CHU de Toulouse
Locations (4):
- France (3):
  - Hôpital du Haut Lévêque, CHU de Bordeaux, Bordeaux
  - Hôpital de la Cavale Blanche, CHU Brest, Brest
  - Hôpital Purpan CIC du CHU de Toulouse, Toulouse
- Centro de Estudos Egas Moniz, Faculdade de Medicina de Lisboa, Lisbon, Portugal